CLINICAL TRIAL: NCT01338558
Title: A Study of Avastin (Bevacizumab) in Combination With mFOLFOX6 in Treatment-Naïve Patients With Metastatic Colorectal Cancer With or Without K-RAS Mutations, and Comparison to Cetuximab
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML25686
Record Dates: First submitted 2011-04-18; First posted 2011-04-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Cetuximab

ARMS (3):
- K-RAS mutated (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: mFOLFOX6
- K-RAS native A (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: mFOLFOX6
- K-RAS native B (Active Comparator)
  Interventions: Drug: cetuximab; Drug: mFOLFOX6

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 5 mg/kg iv on Day 1 of each 2-week cycle until disease progression, unacceptable toxicity or withdrawal of consent
  Arms: K-RAS mutated; K-RAS native A
Drug: cetuximab — 400 mg /m2 iv on Day 1, followed by 250 mg/m2 every week until disease progression, unacceptable toxicity or withdrawal of consent
  Arms: K-RAS native B
Drug: mFOLFOX6 — Standard mFOLFOX6 chemotherapy, 2-week cycles until disease progression, unacceptable toxicity or withdrawal of consent

SUMMARY:
This randomized, open-label study will evaluate the safety and efficacy of Avastin (Bevacizumab) added to standard mFOLFOX6 chemotherapy in treatment-naïve patients with Stage IV metastatic colorectal cancer. According to K-RAS gene mutation status, patients will be assigned or randomized to receive either Avastin 5 mg/kg intravenously (iv) on Day 1 of each 2-week cycle or cetuximab 400 mg/m2 iv on Day 1 followed by 250 mg/m2 iv every week, in addition to mFOLFOX6 every 2 weeks. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >/= 18 years of age
* Histologically confirmed adenocarcinoma of the colon or rectum
* Stage IV metastatic disease with at least one measurable metastatic lesion according to RECIST criteria
* Tumour tissue sample available for assessment of K-RAS and BRAF genes
* Prior radiotherapy must have been completed 4 weeks before randomization
* Adequate bone marrow, kidney and liver function
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Exclusion Criteria:

* Previous chemotherapy for metastatic disease
* Completion of adjuvant treatment for colorectal cancer (Stage I, II and III) in the 12 months preceding randomization
* Prior treatment with bevacizumab, cetuximab or other EGFR inhibitors
* Clinical or radiographic evidence of brain metastases
* Clinically significant cardiovascular disease or disorder
* History of neoplastic disease other than colorectal cancer in the 3 years prior to start of study treatment, except for successfully treated non-invasive carcinomas such as cervical cancer in situ, basal cell carcinoma of the skin or superficial bladder tumours
* HIV, hepatitis B or C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival: native versus mutated K-RAS; tumour assessments according to RECIST criteria | up to 4 years

SECONDARY OUTCOMES:
Overall survival | up to 4 years
Objective response rate | 4 years
Safety: Incidence of adverse events | 4 years
Quality of Life: European Organisation for Research and Treatment of Cancer Quality of Life questionnaire (EORTC QLQ-C30) | up to 4 years
Progression-free survival: comparison of the two treatment regimens in the native K-RAS arms | up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche